CLINICAL TRIAL: NCT04215094
Title: Role of Postoperative Fever, Serum Procalcitonin, C-reactive Protein and White Blood Cell Count in the Diagnosis of Intracranial Infection After Craniotomy
Brief Title: Early Diagnosis of Intracranial Infection After Craniotomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pan Jun (Other)
Responsible Party: Sponsor-Investigator, Pan Jun, PHD, MD,Deputy director of Neurosurgery department, Southern Medical University, China
Organization: Southern Medical University, China (Other)
Other Study IDs: SouthernMUC1
Record Dates: First submitted 2019-11-28; First posted 2020-01-09 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Intracranial; Infection, Psychosis, Acute or Subacute
Keywords: Procalcitonin; C-reactive protein; white blood cell count; intracranial infection
MeSH Terms: conditions — Infections; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- infected group: Intracranial infection were diagnosed according to the Centers for Disease Control (CDC) definitions
  Interventions: Diagnostic Test: postoperative fever, serum procalcitonin, C-reactive protein and white blood cell coun
- non-infected group: the postoperative recovery was uneventful with no infection
  Interventions: Diagnostic Test: postoperative fever, serum procalcitonin, C-reactive protein and white blood cell coun

INTERVENTIONS:
Diagnostic Test: postoperative fever, serum procalcitonin, C-reactive protein and white blood cell coun — All patients in Intracranial Infection group were cured with antibiotic treatment

SUMMARY:
Intracranial infection are serious complications postoperatively in neurosurgical patients. Early identification of these complications is essential to minimize the mortality and moribidy. The aim of this study is observe the postoperative dynamic changes of body temperature (BT), procalcitonin (PCT), C-reactive protein (CRP), and white blood cell (WBC) count, and evaluate whether the use of two or more of these markers may improve the diagnostic accuracy of intracranial infection.

DETAILED DESCRIPTION:
Intracranial infection is a serious complications after neurosurgical operation. Early identification of intracranial infection is important so that, first, optimal treatment is initiated which may improves outcome, second, inappropriate antibiotic treatment and subsequent resistance are prevented, and third, it will promote shorter hospitalization and less cost. In several previous studies, the values of procalcitonin (PCT) and C-reactive protein (CRP) in predicting intracranial infection have been evaluated in neurosurgical patients. However, due to the limited number of studies, the results are not convincing enough and more investigations seems warranted to clarify their dynamic changes in neurosurgical patients without intracranial infection and their role in confirming the suspicion of intracranial infection or excluding intracranial infection from the differential diagnosis.

The aim of the investigator's study is to observe the postoperative dynamic changes of BT, PCT, CRP, and white blood cell (WBC) count, and evaluate whether the use of two or more of these markers may improve the diagnostic accuracy for rational decisions about antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. craniotomy of brain tumor;
2. no clinical manifestations of infection before operation;
3. no other infection such as respiratory tract infection, urinary tract infection and deep vein catheter infection before the definite diagnosis of intracranial infection ;
4. the patients had informed consent to enter the study.

Exclusion Criteria:

1. blood system diseases,respiratory tract infection, urinary tract infection and deep vein catheter infection;
2. malignant tumors with neuroendocrine characteristicsr;
3. aspiration, pancreatitis, etc.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postoperative intracranial infection is one of the most serious complications after neurosurgery. At present, there is no prospective study or recognized effective method for its early diagnosis. It is of great significance for a study about early diagnosis of postoperative intracranial infection,
  In this study, the best diagnostic points of ROC curve will be constructed based on two statistical principles through retrospective study, and then the diagnostic value will be determined through prospective multicenter randomized controlled study. In the research, we will establish quality control system, risk control system and dynamic design to ensure the safety of research subjects and the quality of research results.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-12 (Actual); Primary Completion 2021-07-12 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
the diagnosis of intracranial infection after craniotomy | up to 100 weeks
  Intracranial infection are serious complications postoperatively in neurosurgical patients. Early identification of these complications is essential to minimize the mortality and moribidy. The aim of this study is observe the postoperative dynamic changes of body temperature (BT), procalcitonin (PCT), C-reactive protein (CRP), and white blood cell (WBC) count, and evaluate whether the use of two or more of these markers may improve the diagnostic accuracy of intracranial infection

CONTACTS AND LOCATIONS:
Locations (1):
- Neurosurgery department, Nanfang hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sughrue ME, Bonney PA, Choi L, Teo C. Early Discharge After Surgery for Intra-Axial Brain Tumors. World Neurosurg. 2015 Aug;84(2):505-10. doi: 10.1016/j.wneu.2015.04.019. Epub 2015 Apr 17. PMID 25892244
- [Result] Dubey A, Sung WS, Shaya M, Patwardhan R, Willis B, Smith D, Nanda A. Complications of posterior cranial fossa surgery--an institutional experience of 500 patients. Surg Neurol. 2009 Oct;72(4):369-75. doi: 10.1016/j.surneu.2009.04.001. Epub 2009 Jul 14. PMID 19604553
- [Result] Chidambaram S, Nair MN, Krishnan SS, Cai L, Gu W, Vasudevan MC. Postoperative Central Nervous System Infection After Neurosurgery in a Modernized, Resource-Limited Tertiary Neurosurgical Center in South Asia. World Neurosurg. 2015 Dec;84(6):1668-73. doi: 10.1016/j.wneu.2015.07.006. Epub 2015 Jul 11. PMID 26171888